CLINICAL TRIAL: NCT03356743
Title: Spectrum Analysis of Endobronchial Ultrasound Radiofrequency of Lung Tumors in Ex-vivo Human Lungs
Brief Title: Spectrum Analysis in Ex-vivo Human Lungs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-6177
Record Dates: First submitted 2017-11-13; First posted 2017-11-29 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Lung Cancer
Keywords: lobectomy
MeSH Terms: conditions — Lung Neoplasms | interventions — Spectrum Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ex-Vivo (Experimental)
  Interventions: Device: Spectrum Analysis

INTERVENTIONS:
Device: Spectrum Analysis — The ultrasound probe will be placed on the lung surface in several different directions to obtain the cross section with maximum diameter. Three spectral parameters including midband-fit (dB), intercept (dB), and slope (dB/MHz) will be calculated and compared between the tumor and the lung.

SUMMARY:
This study will analyze spectral features of the radiofrequency of lung tumors in ex-vivo human lungs. The resected specimens will be evaluated using the spectrum analysis to determine the localization rate of the targets. Ultrasound measurement and images will be used for correlation of TS mode image findings with pathology by using HE and IHC slides of lung tumor and lymph node.

ELIGIBILITY:
Inclusion Criteria:

* Any patients scheduled for lobectomy of anatomical segmental resection for malignant lung tumors.
* 18 years of age or older

Exclusion Criteria:

* Any patients with inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
To analyze the relationship of three spectral features of the radiofrequency of lung tumors in ex-vivo human lungs. | Within an hour after resection.
  From obtained ultrasound images, a linear regression line is quantified, and three ultrasonic spectral parameters including Midband-fit, Intercept, and Slope are calculated.

SECONDARY OUTCOMES:
To find the correlation of TS mode image findings with pathology by using lung tumor and lymph node samples. | Within an hour after resection
  After evaluation, the actual tumor size and histological diagnosis will be determined. Differences between US image and pathological morphology will be determined by using HE and Immunohistochemistry (IHC) slides of lung tumor, the investigators will evaluate comparison of nucleus size in each tissue and the spectral parameters in each region of interest.
To clarify the feasibility of using the conventional EBUS scope to visualize solitary pulmonary nodules in an ex-vivo human lung. | Within an hour after resection
  The bronchial stump of the specimen will be opened and a small sized endotracheal tube will be inserted to inflate and deflate the lung. After inflation of the lung, visualization of the tumor will be evaluated to see the difference in ultrasound images between deflated and inflated lung.

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Plan on sharing data at the time of manuscript publication.